CLINICAL TRIAL: NCT00822809
Title: Two-arm, Randomized, Open-label, Phase IIIb Study Investigating the Safety of a 3 Hour i.p. Infusion of Catumaxomab With and Without Prednisolone Premedication in Patients With Malignant Ascites Due to Epithelial Cancer
Brief Title: CASIMAS: Catumaxomab Safety Phase IIIb Study With Intraperitoneal Infusion in Patients With Malignant Ascites Due to Epithelial Cancers
Acronym: CASIMAS
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Neovii Biotech (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: IP-CAT-AC-03
Record Dates: First submitted 2008-12-23; First posted 2009-01-14 (Estimated); Last update posted 2012-10-03 (Estimated); Status verified 2012-08

CONDITIONS: Cancer; Neoplasms; Carcinoma; Malignant Ascites
Keywords: Cancer; Neoplasms; Carcinoma; Malignant Ascites; Drug therapy; Antineoplastic Protocols; Immunotherapy; Phase III; trifunctional antibody; monoclonal antibody; EpCAM
MeSH Terms: conditions — Neoplasms; Carcinoma | interventions — catumaxomab; Prednisolone

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- A (Experimental): Patients will receive premedication of 25 mg (i.v.) prednisolone 30 minutes prior start of infusion of catumaxomab.
  Catumaxomab will be infused i.p. with 3 hour constant rate infusions via an indwelling catheter.
  Interventions: Drug: Catumaxomab; Drug: Prednisolone
- B (Other): Catumaxomab will be administered in a dosage identical to Arm A but without the prednisolone premedication.
  Interventions: Drug: Catumaxomab

INTERVENTIONS:
Drug: Catumaxomab — Catumaxomab will be infused 4 times within 11 days as follows:
  10 µg on day 0, 20 µg on day 3, 50 µg on day 7, 150 µg on day 10
Drug: Prednisolone — 25 mg premedication
  Arms: A

SUMMARY:
This is a randomized phase IIIb study investigating the treatment of malignant ascites due to epithelial cancer (carcinomas) with the trifunctional antibody catumaxomab. In order to make the catumaxomab treatment more convenient for the patient and the hospital praxis the tolerability of 3 hour infusions of catumaxomab with and without premedication of prednisolone is evaluated.

A total of 208 patients with malignant ascites due to epithelial cancer will be allocated to two treatment groups in a 1:1 ratio.

DETAILED DESCRIPTION:
Safety data of the completed pivotal phase II/III trial, IP-REM-AC-01, in which catumaxomab was administered as 6 hour i.p. infusion showed that most reported AEs were cytokine release-related symptoms such as fever, nausea, and vomiting (based on the pharmacodynamic mode of action of catumaxomab) and abdominal pain. In order to make the catumaxomab treatment more convenient for the patient and the hospital praxis the current trial was designed to determine whether tolerability of the 3 hour infusion of catumaxomab with and without premedication of prednisolone. Prednisolone was chosen as additional premedication with the objective to reduce cytokine release related symptoms which might change with the switch from 6 to 3 h infusion time.

ELIGIBILITY:
Key Inclusion Criteria:

1. Patients with malignant ascites requiring therapeutic ascites puncture
2. Histological confirmed diagnosis of epithelial cancer
3. Patients where standard therapy is not available or no longer feasible
4. Karnofsky index ≥60 %
5. Life expectancy >12 weeks

Key Exclusion Criteria:

1. Concomitant treatment with other investigational product, chemo-, or radiotherapy
2. Recent exposure to an investigational product
3. Known or suspected hypersensitivity to catumaxomab or similar antibodies
4. Inadequate respiratory, renal or hepatic function
5. Inadequate blood count (platelets, neutrophils)
6. Required entirely parenteral nutrition
7. Patients with ileus or subileus within the last 30 days
8. Liver metastases with volume >70 % of liver tissue
9. Known portal vein obstruction
10. Known Brain metastases
11. Acute or chronic infection
12. Not sufficiently recovered from previous treatment (toxicity present) based on laboratory values and general status
13. Albumin lower than 3 g/dL or total protein < 6g/dL

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 230 (Actual)
Dates: Start 2008-12; Primary Completion 2010-11 (Actual); Study Completion 2011-04 (Actual)

PRIMARY OUTCOMES:
Influence of prednisolone on the safety of 3 hours i.p. infusion of catumaxomab measured by a composite safety score | 6 months
Puncture-free survival defined as the time from clock start to first need for therapeutic ascites puncture or death, whichever occurs first. | 6 months

SECONDARY OUTCOMES:
Safety measured by • Incidence of all AEs, • Changes in clinically relevant laboratory values (hematology, clinical chemistry, coagulation, and urinalysis), • Physical examination, • Vital signs. | 6 months
Time to next ascites puncture, number of ascites punctures until end of lifetime, overall survival, anti-cancer treatment | 6 months
immune monitoring | 6 months

CONTACTS AND LOCATIONS:
Overall Officials: Florian Lordick, PD Dr. med., Principal Investigator — Med. Klinik III, Städtisches Klinikum Braunschweig gGmbH, Celler STr. 38, 38114 Braunschweig
Locations (4):
- Study Site, Several, France
- Study site, Several, Germany
- Study Site, Several, Italy
- Study Site, Several, Spain

REFERENCES:
- [Background] Lordick F, Ott K, Weitz J, Jager D. The evolving role of catumaxomab in gastric cancer. Expert Opin Biol Ther. 2008 Sep;8(9):1407-15. doi: 10.1517/14712598.8.9.1407. PMID 18694358
- [Background] Burges A, Wimberger P, Kumper C, Gorbounova V, Sommer H, Schmalfeldt B, Pfisterer J, Lichinitser M, Makhson A, Moiseyenko V, Lahr A, Schulze E, Jager M, Strohlein MA, Heiss MM, Gottwald T, Lindhofer H, Kimmig R. Effective relief of malignant ascites in patients with advanced ovarian cancer by a trifunctional anti-EpCAM x anti-CD3 antibody: a phase I/II study. Clin Cancer Res. 2007 Jul 1;13(13):3899-905. doi: 10.1158/1078-0432.CCR-06-2769. PMID 17606723
- [Background] Shen J, Zhu Z. Catumaxomab, a rat/murine hybrid trifunctional bispecific monoclonal antibody for the treatment of cancer. Curr Opin Mol Ther. 2008 Jun;10(3):273-84. PMID 18535935
- [Derived] Fossati M, Buzzonetti A, Monego G, Catzola V, Scambia G, Fattorossi A, Battaglia A. Immunological changes in the ascites of cancer patients after intraperitoneal administration of the bispecific antibody catumaxomab (anti-EpCAMxanti-CD3). Gynecol Oncol. 2015 Aug;138(2):343-51. doi: 10.1016/j.ygyno.2015.06.003. Epub 2015 Jun 3. PMID 26049121